CLINICAL TRIAL: NCT00174317
Title: Clinical Protocol For A Multicentre, Double-Blind, Randomised, Parallel Group Study To Compare The Efficacy and Tolerability Of Celecoxib Vs. Diclofenac In The Treatment Of Subjects With Osteoarthritis Of The Hip Requiring Joint Replacement Therapy
Brief Title: Celecoxib Versus Diclofenac In The Treatment Of Osteoarthritis Of The Hip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COXA-0508-261
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2005-12

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Celecoxib; Diclofenac

INTERVENTIONS:
Drug: Celecoxib
Drug: Diclofenac

SUMMARY:
To determine if celecoxib 200 mg once daily is as effective as diclofenac 50 mg three times daily in the treatment of pain symptoms associated with osteoarthritis of the hip

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with osteoarthritis of hip and requiring joint replacement
* Eligible for chronic therapy with an NSAID

Exclusion Criteria:

* Hip surgery anticipated within 8 calendar weeks after first visit
* Active gastrointestinal disease or recent diagnosis of gastrointestinal ulceration (within 60 days of first visit)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-08; Study Completion 2005-02

PRIMARY OUTCOMES:
Change in patient assessment of arthritis pain on walking VAS (Visual Analog Scale) as measured on a 0-100 mm scale at week 6 compared to baseline

SECONDARY OUTCOMES:
Change in patient assessment of arthritis pain on walking VAS (Visual Analog Scale) as measured on a 0-100 mm scale at week 12 compared to baseline.
Change in patients global assessment of arthritis between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United Kingdom (42):
  - Pfizer Investigational Site, Aston Clinton, Bucks
  - Pfizer Investigational Site, Ely, Cambs
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Lancaster, England
  - Pfizer Investigational Site, Sheffield, England
  - Pfizer Investigational Site, Newport, Gwent
  - Pfizer Investigational Site, Chingford, London
  - Pfizer Investigational Site, Harrow, MIDDLESEX
  - Pfizer Investigational Site, Greenisland, Carrickfergus, Northern Ireland
  - Pfizer Investigational Site, Oxford, Oxon
  - Pfizer Investigational Site, Greenock, Renfrewshire
  - Pfizer Investigational Site, Barry, South Glamorgan
  - Pfizer Investigational Site, Barnsley, South Yorkshire
  - Pfizer Investigational Site, Ashford, Surrey
  - Pfizer Investigational Site, Newcastle upon Tyne, Tyne & Wear
  - Pfizer Investigational Site, Trowbridge, Wiltshire
  - Pfizer Investigational Site, Aberdeen
  - Pfizer Investigational Site, Amersham
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Bradford
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Carshalton
  - Pfizer Investigational Site, Chertsey
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Lancaster
  - Pfizer Investigational Site, Leystonstone, London
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Northampton
  - Pfizer Investigational Site, Norwich
  - Pfizer Investigational Site, Nuneaton
  - Pfizer Investigational Site, Peterborough
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Truro
  - Pfizer Investigational Site, Wansford
  - Pfizer Investigational Site, Watford
  - Pfizer Investigational Site, Westbury
  - Pfizer Investigational Site, Wigan